CLINICAL TRIAL: NCT07296497
Title: A Randomized, Multicenter, Single-blind, Sham-controlled Clinical Trial on the Efficacy and Safety of Acupuncture in the Treatment of Refractory Rosacea.
Brief Title: Acupuncture for Refractory Rosacea: A Study on Its Effectiveness and Safety
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 202507085-2
Record Dates: First submitted 2025-11-24; First posted 2025-12-22 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-10

CONDITIONS: Rosacea
Keywords: rosacea; acupuncture
MeSH Terms: conditions — Rosacea | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupuncture group (Experimental)
  Interventions: Device: Acupuncture
- sham acupuncture group (Sham Comparator)
  Interventions: Procedure: Sham Acupuncture

INTERVENTIONS:
Device: Acupuncture — The acupuncture sites are primarily located on the face, neck, and proximal limbs along major blood vessels. The specific acupoints include Jiquan (HT1), Yinlian (LR11), Weizhong (BL40), Chize (LU5), and facial Ashi points. The needles are inserted to a depth of 2-3 mm, retained, and stimulated with continuous waves at a frequency of 1 Hz for 20 minutes. Electrical stimulation is not applied to the facial Ashi points, where needles are retained only. The treatment course lasts for 8 weeks, with two sessions per week, for a total of 16 sessions.
  Arms: acupuncture group
Procedure: Sham Acupuncture — Use blunt-tipped acupuncture needles to deliver sham stimulation. The blunt needles do not penetrate the skin. The treatment sites, needle retention time, and electrical stimulation frequency are identical to those in the acupuncture group. The treatment duration and frequency are also the same as in the acupuncture group.
  Arms: sham acupuncture group

SUMMARY:
This study is a randomized, multicenter, sham-controlled clinical trial designed to evaluate the efficacy and safety of acupuncture for patients with refractory rosacea. A total of 104 participants will be enrolled and randomly assigned in a 1:1 ratio to the acupuncture group or the sham acupuncture group (52 participants in each group, regardless of sex). The primary aim is to determine whether acupuncture can effectively alleviate facial erythema and flushing episodes compared with sham stimulation.

DETAILED DESCRIPTION:
Participants in the acupuncture group will receive electroacupuncture treatment using continuous waves at a frequency of 1 Hz, delivering microcurrent intensity comparable to human bioelectric levels for 20 minutes per session. Participants in the sham group will receive noninvasive stimulation with blunt-tipped needles that do not penetrate the skin. The study duration is 17 weeks in total, consisting of a 1-week baseline observation period, an 8-week treatment phase (16 treatment sessions in total), and an 8-week follow-up phase. Five in-person assessment visits will be conducted at weeks 0, 4, 8, and 12, followed by an online follow-up at week 16. The study will assess improvements in rosacea symptoms and monitor treatment safety throughout the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with refractory rosacea, defined as those who have received at least 12 weeks of conventional oral medication (such as doxycycline), with or without other treatments (e.g., topical medications or intense pulsed light [IPL] therapy), but remain treatment-resistant - characterized by no improvement of erythema by at least one CEA grade, persistent erythema ≥ grade 3, or recurrent flushing that affects quality of life (DLQI indicating at least a moderate impact); or patients who experience frequent relapses during the 12-week treatment period;
2. Age between 18 and 65 years, inclusive, with no restriction on sex;
3. Individuals who fully understand the purpose and significance of the study, voluntarily agree to participate, sign the informed consent form (ICF), and are willing to comply with all study procedures and follow-up requirements.

Exclusion Criteria:

1. Women who are pregnant, breastfeeding, or planning to become pregnant in the near future;
2. Patients with diabetes mellitus or moderate to severe systemic diseases affecting the liver, kidney, lung, or hematologic system;
3. Patients with depression or other psychiatric disorders;
4. Individuals with severe abnormal reactions to acupuncture (e.g., syncope during acupuncture, allergy to acupuncture needles);
5. Patients with rosacea accompanied by nasal hypertrophy or other facial dermatoses (such as seborrheic dermatitis, eczema) or facial manifestations of other systemic diseases (such as dermatomyositis, systemic lupus erythematosus);
6. Individuals with a bleeding tendency or coagulation disorders, or with skin damage, infection, or other lesions at the acupuncture sites;
7. Patients who discontinued oral antibiotics less than 1 month prior to enrollment; discontinued non-antibiotic oral medications less than 15 days prior (or isotretinoin less than 3 months prior); or discontinued topical medications less than 1 week prior;
8. Patients who are expected to be unable to comply with follow-up requirements;
9. Individuals who have participated in any other clinical trial within 1 month before screening (defined as having signed an informed consent form and received an investigational drug/device/placebo);
10. Any other condition that, in the opinion of the investigator, makes the participant unsuitable for enrollment.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-12-24 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
proportion of successful treatment for rosacea erythema | week0，4，8，12
  The treatment is defined as successful when the Clinician's Erythema Assessment (CEA) score is ≤ 1 or has decreased by 2 points from baseline.

SECONDARY OUTCOMES:
improvement in severity of rosacea flushing | week0，4，8，12
  This outcome is evaluated using the Rosacea Clinical Severity Assessment Scale - Patient Version (RCSAS-P), a patient-reported questionnaire capturing daily symptom burden. Patients score subjective symptoms-including facial flushing, erythema intensity, burning/stinging sensations, warmth, and overall discomfort-on structured rating items. The scale reflects symptom severity from the patient's perspective and complements clinician assessments.
improvement in burning sensation severity in rosacea | week0，4，8，12
  This outcome is evaluated using the Rosacea Clinical Severity Assessment Scale - Patient Version (RCSAS-P), a patient-reported questionnaire capturing daily symptom burden. Patients score subjective symptoms-including facial flushing, erythema intensity, burning/stinging sensations, warmth, and overall discomfort-on structured rating items. The scale reflects symptom severity from the patient's perspective and complements clinician assessments.
improvement in degree of telangiectasia in rosacea | week0，4，8，12
  This outcome is evaluated using the Rosacea Clinical Severity Assessment Scale - Patient Version (RCSAS-P), a patient-reported questionnaire capturing daily symptom burden. Patients score subjective symptoms-including facial flushing, erythema intensity, burning/stinging sensations, warmth, and overall discomfort-on structured rating items. The scale reflects symptom severity from the patient's perspective and complements clinician assessments.
Pittsburgh Sleep Quality Index (PSQI) | week0，4，8，12
Rosacea-Specific Quality of Life Questionnaire (RosQoL) | week0，4，8，12
improvement in the number/frequency of weekly flushing episodes in rosacea | week0，4，8，12
  This outcome is evaluated using the Rosacea Diary, a structured patient-reported daily log designed to document symptom fluctuations. Participants record the presence, frequency, and severity of flushing episodes, as well as associated erythema, burning, stinging, and discomfort. The diary captures day-to-day variability and provides quantitative data on weekly flushing patterns and symptom burden.
Number of participants with treatment-related adverse events as assessed by the Rosacea Treatment-Related Adverse Event Recording Form (RTAERF) | week0，4，8，12
  Treatment-related adverse events (AEs) will be collected using the Rosacea Treatment-Related Adverse Event Recording Form (RTAERF), an investigator-developed safety assessment tool. The form captures all local and systemic AEs, including onset, duration, severity, relationship to the intervention, and outcome. AEs will be summarized as the number and proportion of participants experiencing at least one treatment-related AE during the study period. Serious adverse events (SAEs) will also be documented and reported separately.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: No
Only aggregated statistical results will be shared through academic publication. Individual participant data will not be shared due to confidentiality and privacy protection requirements.